CLINICAL TRIAL: NCT01916057
Title: Multicenter Prospective Pilot Study Investigating Pathophysiology, Diagnostic and Therapeutic Strategies of Hepatosplenic Candidiasis
Brief Title: Hepatosplenic CANdidiasis : PETscan and Immune Response Analysis
Acronym: CANHPARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Lausanne Hospitals (Other); University Hospital, Lille (Other); Institut Pasteur (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120115; AOM12047
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Invasive Fungal Disease; Chronic Disseminated Candidiasis; Hematological Malignancies; Hematopoietic Stem Cell Transplantation; Neutropenia
Keywords: Positron-Emission Tomography Scan; Fluorodeoxyglucose F18; Magnetic Resonance Imaging; Enzyme-Linked Immunospot Assay; Immune Reconstitution Inflammatory Syndrome; Real-Time Polymerase Chain Reaction; beta-1,3-D-glucan; Candida spp.; Genetic Susceptibility; Genotype
MeSH Terms: conditions — Invasive Fungal Infections; Hematologic Neoplasms; Neutropenia; Immune Reconstitution Inflammatory Syndrome; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-FDG PET Scan (Experimental): 18F-FDG PET Scan at Day 0 and M3
  Interventions: Device: 18F-FDG PET Scan

INTERVENTIONS:
Device: 18F-FDG PET Scan — to determine whether F18 fluorodeoxyglucose (18F-FDG) positron-emission tomography scan (PET scan) is useful for the therapy strategy of hepatosplenic candidiasis.

SUMMARY:
The purpose of this study is to determine whether F18 fluorodeoxyglucose (18F-FDG) positron-emission tomography scan (PET scan) is useful for the therapy strategy of hepatosplenic candidiasis.

DETAILED DESCRIPTION:
Chronic disseminated candidiasis, often referred to as hepatosplenic candidiasis (HSC), is an infection due to Candida spp. that mainly involves the liver and spleen. HSC occurs mostly in patients with profound and prolonged neutropenia, which is more often seen in patients with hematologic malignancies. Despite an appropriate antifungal prophylaxis, the incidence of HSC in France might be closed to 5% in patients suffering from acute leukemia. Early and adequate diagnosis and treatment of HSC are crucial, as treatment delays can negatively affect the prognosis of the underlying condition. Current guidelines recommend a 6-month duration treatment. Prolonged treatments up to 6 months are frequent, leading to antifungal toxicity and cost increase. Preliminary study by our team has already assessed F18 fluorodeoxyglucose (18F-FDG) positron-emission tomography scan (PET scan) as a diagnostic tool for HSC. 18F-FDG PET scan could be helpful in the diagnosis, follow-up and therapy strategy of HSC, helping to stop antifungal treatment. Other molecular, immunological and serological tools have to be developed in order to avoid hepatic biopsies. Actually, mycological evidence of infection is found in only 20% of the cases. The pathogenesis of HSC is also not well understood, but it is believed that it may be due to an unbalanced adaptive immune response that leads to an exacerbated inflammatory reaction, resulting in an Immune Reconstitution Inflammatory Syndrome (IRIS). In that context, a better understanding of the disease pathophysiology and of the potential genetic susceptibility could have an impact on therapy strategy. For example, new approaches such as the use of adjuvant high-dose corticosteroids have been shown beneficial. This study is the first step to improve HSC diagnosis and therapy strategy.

ELIGIBILITY:
Patients' inclusion criteria:

* Adults aged ≥18 years-old
* Hospitalized for hematological malignancy or hematopoietic stem cell transplantation
* Recent (>2months), prolonged (>10 days), profound (>100 PMN/mm3), feverish neutropenia
* Suspected hepatosplenic candidiasis (typical small nodular lesions on abdominal RMI or CT)

Patients' exclusion criteria:

- hepatosplenic lesions of other proven origin

Patients' non-inclusion criteria:

* Life expectancy >3 months
* Pregnancy
* HIV infection
* Hepatic biopsy within 3 weeks before 18F-FDG PET scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Global response to therapy | at month 3
  Clinical assessment (no fever) and PET scan assessment (intensity of liver and/or spleen lesions)

SECONDARY OUTCOMES:
18F-FDG PET scan and RMI usefulness in initial diagnosis | at month 3
  Comparison between Day 0 and Month 3 exams
Serological and molecular mycological tools assessment | at day 0
  Measurement of beta-1,3-D-glucans, mannan/anti-mannan, anti-Saccharomyces cerevisiae antibodies in comparison with controls.
  Assessment of a new real-time PCR on serum and hepatic tissue
Serological and molecular mycological tools assessment | at Month 3
  Measurement of beta-1,3-D-glucans, mannan/anti-mannan, anti-Saccharomyces cerevisiae antibodies in comparison with controls.
  Assessment of a new real-time PCR on serum and hepatic tissue
Serological and molecular mycological tools assessment | at Month 6
  Measurement of beta-1,3-D-glucans, mannan/anti-mannan, anti-Saccharomyces cerevisiae antibodies in comparison with controls.
  Assessment of a new real-time PCR on serum and hepatic tissue
Inflammatory cells and mediators | at day 0
  Measurement of cytokines and lymphocytes populations on serum and hepatic tissue in comparison with controls
Inflammatory cells and mediators | at month 3
  Measurement of cytokines and lymphocytes populations on serum and hepatic tissue in comparison with controls
Inflammatory cells and mediators | at month 6
  Measurement of cytokines and lymphocytes populations on serum and hepatic tissue in comparison with controls
Genetic susceptibility | at day 0
  Search for susceptibility genes to candidiasis in comparison with controls

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - Centre d'Infectiologie Necker-Pasteur, IHU Imagine - Hôpital Necker-Enfants Malades,, Paris, France

REFERENCES:
- [Background] Rammaert B, Maunoury C, Rabeony T, Correas JM, Elie C, Alfandari S, Berger P, Rubio MT, Braun T, Bakouboula P, Candon S, Montravers F, Lortholary O. Does 18F-FDG PET/CT add value to conventional imaging in clinical assessment of chronic disseminated candidiasis? Front Med (Lausanne). 2022 Dec 20;9:1026067. doi: 10.3389/fmed.2022.1026067. eCollection 2022. PMID 36606049
- [Background] Candon S, Rammaert B, Foray AP, Moreira B, Gallego Hernanz MP, Chatenoud L, Lortholary O. Chronic Disseminated Candidiasis During Hematological Malignancies: An Immune Reconstitution Inflammatory Syndrome With Expansion of Pathogen-Specific T Helper Type 1 Cells. J Infect Dis. 2020 May 11;221(11):1907-1916. doi: 10.1093/infdis/jiz688. PMID 31879764